CLINICAL TRIAL: NCT02710266
Title: Evaluation of the Effect of Gabexate Mesilate in the Hepatocyte Protection After Liver Resection
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was closed earlier than planned because targeted participant recruitment is not smooth.
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2011-0936
Record Dates: First submitted 2016-02-01; First posted 2016-03-16 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Liver Disease
Keywords: Synthetic Protease Inhibitor; Hepatectomy; Postoperative Complications
MeSH Terms: conditions — Liver Diseases; Postoperative Complications | interventions — Hepatectomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo group (Placebo Comparator): hepatectomy without Gabexate Mesilate
  Interventions: Drug: hepatectomy with dextrose water
- Preoperative Gabexate Mesilate group (Experimental): Gabexate Mesilate administered from the preoperative day
  Interventions: Drug: Preoperative Gabexate Mesilate group
- Intraoperative Gabexate Mesilate group (Experimental): Gabexate Mesilate administered from the operative day
  Interventions: Drug: Intraoperative Gabexate Mesilate group

INTERVENTIONS:
Drug: Preoperative Gabexate Mesilate group — Gabexate Mesilate is administered from the preoperative day and continued for 5 days. 300mg of Gabexate Mesilate is mixed with 500cc of 5% dextrose water and administered at 40cc/hr for 12 hours each day.
  Arms: Preoperative Gabexate Mesilate group
Drug: Intraoperative Gabexate Mesilate group — Gabexate Mesilate is administered from the operative day and continued for 5 days. 300mg of Gabexate Mesilate is mixed with 500cc of 5% dextrose water and administered at 40cc/hr for 12 hours each day.
  Arms: Intraoperative Gabexate Mesilate group
Drug: hepatectomy with dextrose water — Gabexate Mesilate is not administered. As placebo, 500cc of 5% dextrose water is administered at 40cc/hr for 12 hours
  Arms: Placebo group

SUMMARY:
Liver resection have been a primary treatment option for lesions found in the liver. With improvements in surgical technique and perioperative patient management, morbidity and mortality related to liver resection have been greatly reduced. However, many patients with hepatocellular carcinoma have underlying liver disease. Severity of underlying liver disease plays an important role in decision making of resection extent. Therefore, liver failure and decreased liver function following liver resection still remains to be an critical issue.

Postresection liver failure is generally defined by serum total bilirubin greater than 3mg/dL and prothrombin time of less than 50% of normal (INR >1.7). Pathophysiology of postresection liver failure is not yet well known. However, sepsis after liver resection, small-for-size syndrome (SFSS), and ischemia/reperfusion injury are known to have important roles in persistant liver injury after resection.

After a liver resection, kupffer cells are drastically decreased and innate immunity of the patient is also damaged. This process causes the patient to be vulnerable to infection. In addition, with continuous endotoxin secretion, dysfunction in kupffer cells are triggered and liver regeneration is affected.

Complex mechanisms leading to dysfunctional kupffer cells and apoptosis and necrosis of hepatocytes are mediated by neutrophils, complement, reactive oxygen species, and acute inflammatory cytokines.

Recent studies have reported on many promising effects of the synthetic protease inhibitor, such as Gabexate mesilate. These include antioxidant effect, inhibition of acute inflammatory cytokine reaction, and anticoagulatory property. Based on these effects, synthetic protease inhibitor have gained attention in the role of hepatocyte protection after liver resection.

Currently, there is a report on the hepatocyte protective effects of Gabexate Mesilate on ischemia/reperfusion injury caused by the Pringle maneuver. However, with the advances in surgical technique and equipment, many surgeons now perform liver resection without Pringle maneuver. Therefore, this study was designed to determine effects of Gabexate Mesilate in the liver resection performed without Pringle maneuver.

ELIGIBILITY:
Inclusion Criteria:

* All liver tumors that require resection of more than two segments of the liver.
* Age ≥20 and ≤80
* General performance status: the Karnofsky score> 70% or ECOG 0-1

Exclusion Criteria:

* Hepatic duct reconstruction was performed
* ASA (American society of anesthesiologists' physical status classification) score: ≥3
* Patients with drug or alcohol addiction
* Patients showing low compliance
* Patients who not want to involve the clinical trial
* Patients who are unable to read or understand the informed consent, sign a consent form (eg, mental retardation, blindness, illiteracy, foreign, etc.)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-02-24 (Actual); Primary Completion 2017-02-25 (Actual); Study Completion 2017-02-25 (Actual)

PRIMARY OUTCOMES:
Postoperative complications | Within the first 30 days after surgery

SECONDARY OUTCOMES:
Liver function recovery time | 4 weeks
length of hospitalization | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim YI, Fujita S, Hwang YJ, Chun JM, Song KE, Chun BY. Successful intermittent application of the Pringle maneuver for 30 minutes during human hepatectomy: a clinical randomized study with use of a protease inhibitor. Hepatogastroenterology. 2007 Oct-Nov;54(79):2055-60. PMID 18251159